CLINICAL TRIAL: NCT05611099
Title: Assessment of the Stability, Robustness and Usability of the Dreem 3 System for EEG Sleep Monitoring in the Home Setting, in an Insomnia Population.
Brief Title: Robustness and Usability of the Dreem 3 System for at Home Sleep Monitoring in an Insomnia Population.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dreem (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LIVIE-1
Record Dates: First submitted 2022-11-01; First posted 2022-11-09 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Insomnia, Secondary; Sleep Disturbance; Sleep; Sleep Initiation and Maintenance Disorders
Keywords: Polysomnography; Sleep assessment; Dreem; EEG; dry EEG; Accuracy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Parasomnias

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Dreem + WatchPAT One (Experimental): Single arm of 15 subjects wearing simultaneously the Dreem 3 + WatchPAT One devices for 3 nights, and then undergoing an end of study usability questionnaire.
  Interventions: Device: Dreem 3 System vs WatchPAT One; Other: Usability Questionnaire

INTERVENTIONS:
Device: Dreem 3 System vs WatchPAT One — Dreem 3 System and WatchPAT One will be worn simultaneously during 3 nights by each study participant, in order to compare the TST automatically outputted by both devices.
Other: Usability Questionnaire — After having undergone the 3 nights of measurement, an end of Study Questionnaire will be performed on a separate day to obtain Usability feedback from participants who have undergone simultaneous recordings with the Dreem 3 + WatchPAT devices.

SUMMARY:
There is an unmet medical need for monitoring sleep for multiple nights in a patient's home, without the inconvenience of traveling and staying overnight in a medical center, and without the need for a technician to set up a polysomnography (PSG) device at the patient's home. Several disorders, and particularly sleep disorders, are associated with insomnia symptoms, and longitudinal sleep assessment may support a better understanding and management of these patients, who currently seldom access sleep lab PSG.

On one hand, this study aims at demonstrating whether the final device's user interface supports safe and effective use when being used at home over multiple nights.

On the other, the study aims at confirming that stable and consistent data are measured in the device's actual use, for the records to be clinically usable in daily practice.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be ≥ 22 and ≤ 70 years old inclusive, including:

  * 8 subjects under 55 years old.
  * 7 subjects over 55 years old.
* Subjects who are under the care of a sleep clinician for experiencing insomnia symptoms.
* Subjects have wifi connection at their home.
* Subjects have a smartphone where they can install the Alfin App.
* Subjects agree to not having abnormal drugs or alcohol consumption 24 hours before the start of the measurement, and during the 3 days of measurement.
* Able to read, understand and sign an informed consent form.

Exclusion Criteria:

* Under 22 and above 70 years old inclusive.
* BMI ≥ 40.
* Obstructive sleep apnea diagnosis with ongoing CPAP therapy.
* Abnormal drugs or alcohol use during the measurement part of the study.
* Head circumference < 53 cm or device fitting issues as determined during training.
* Not able to read, understand and sign an informed consent form.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-11-05 (Actual)

PRIMARY OUTCOMES:
TST Correlation | 3 nights
  Pearson's Correlation between the total time (in minutes) the subject spends asleep (TST) as automatically determined by the Dreem 3S compared to the TST automatically determined by the WatchPAT One (WP1) device on the same night.
Dreem 3 System usability | 1 day
  As determined by the System Usability Scale. The System Usability Scale establishes a score (the SUS score), between 0 and 100. A score of 68 indicates average performance of a system. A score > 68 indicated the system's usability is above average.

SECONDARY OUTCOMES:
ΔTST Correlation | 3 nights
  Pearson's correlation on Dreem 3S and WP1 intra-subject, inter-nights TST differences.

OTHER OUTCOMES:
Detailed Usability Questionnaire | 1 day
  Quantitative feedback on the critical tasks of the Dreem 3 System over multiple nights in a home environment. Questions are graded from "Strongly Disagree" to "Strongly Agree", where strongly agree means the subject understands how to interact with the different subparts of the Dreem 3S and experiences no usability issue.
Usability Interview | 1 day
  Qualitative information regarding the perceptions, opinions, beliefs and attitudes of individuals on the overall subjective experience of the Dreem 3 System over multiple nights in a home environment.

CONTACTS AND LOCATIONS:
Locations (1):
- Dreem Health, Encinitas, California, United States

IPD SHARING:
Plan to Share IPD: No